CLINICAL TRIAL: NCT03064113
Title: A Phase 2, Randomized, Double-Blind, Crossover Study to Examine the Pharmacodynamics, Safety and Tolerability, and Pharmacokinetics of Single Doses of TD-4208 in Subjects Diagnosed With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of TD-4208 on FEV1 in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0059; ACTRN12611000482965 (Registry Identifier: ANZCTR); U1111-1120-8290 (Other: Universal Trial Number)
Record Dates: First submitted 2017-01-20; First posted 2017-02-24 (Actual); Results first posted 2019-11-14 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease, COPD
Keywords: Chronic Obstructive Pulmonary Disease, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental): Period 1 = Placebo; Period 2 = TD-4208 700 μg; Period 3 = TD-4208 350 μg; Period 4 = Ipratropium 500 μg
  Interventions: Drug: Placebo; Drug: TD-4208 700 μg; Drug: TD-4208 350 μg; Drug: Ipratropium 500 μg
- Sequence 2 (Experimental): Period 1 = TD-4208 700 μg; Period 2 = Ipratropium 500 μg; Period 3 = Placebo; Period 4 = TD-4208 350 μg
  Interventions: Drug: Placebo; Drug: TD-4208 700 μg; Drug: TD-4208 350 μg; Drug: Ipratropium 500 μg
- Sequence 3 (Experimental): Period 1 = TD-4208 350 μg; Period 2 = Placebo; Period 3 = Ipratropium 500 μg; Period 4 = TD-4208 700 μg
  Interventions: Drug: Placebo; Drug: TD-4208 700 μg; Drug: TD-4208 350 μg; Drug: Ipratropium 500 μg
- Sequence 4 (Experimental): Period 1 = Ipratropium 500 μg; Period 2 = TD-4208 350 μg; Period 3 = TD-4208 700 μg; Period 4 = Placebo
  Interventions: Drug: Placebo; Drug: TD-4208 700 μg; Drug: TD-4208 350 μg; Drug: Ipratropium 500 μg

INTERVENTIONS:
Drug: Placebo
Drug: TD-4208 700 μg
  Other Names: Revefenacin
Drug: TD-4208 350 μg
  Other Names: Revefenacin
Drug: Ipratropium 500 μg

SUMMARY:
Thirty-two subjects diagnosed with COPD were enrolled, received each study treatment and completed the follow-up assessments. During each of the four study periods, subjects were admitted to the clinic on Day -1 and housed overnight until after the last spirometry measurement. Serial pulmonary function tests were performed and PK (pharmacokinetics) samples collected up to 25 hours. Subjects were discharged from the clinic on Day 2 after evaluations.

DETAILED DESCRIPTION:
Subjects were assigned to one of the 4-treatment sequence groups presented in the table above according to a randomization schedule supplied by the Sponsor before study initiation. The randomization scheme did not include assignments for replacement subjects.

Subjects reported to their respective clinical research unit (CRU) on Admission/Day -1 for pre-randomization procedures and confirmation of eligibility (and continued eligibility for Periods 2 to 4). The unblinded pharmacist prepared and dispensed the nebulizers, according to the randomization schedule for each of the 4 periods. Dosing occurred in the morning, generally between 7 am and 9 am. For Periods 2 to 4, dosing occurred within ±30 minutes of the dosing time established in Period 1.

Study drug was administered in the respective CRU under the supervision of study personnel. Single doses of TD-4208, ipratropium bromide, and placebo were administered in the clinical research unit (CRU) under the supervision of study personnel. Care was taken to avoid eye contact with study drugs. Residual drug solution remaining in the nebulizer (ie, in mL) was measured and recorded.

The investigator or designee was responsible for maintaining accountability records for all study drug(s) in accordance with applicable government regulations and study procedures.

The accountability record included entries for receipt, distribution or dispensing, and destruction of the material(s). Unused and expired study drugs were to be disposed of in accordance with written instructions from the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate stable Chronic Obstructive Pulmonary.
* Disease with FEV1/FVC <0.7 at screening.
* Woman of non-childbearing potential.
* Female participants of childbearing potential must test negative for pregnancy and must be using a highly effective method of birth control during the study and for at least 1 month after completion of study dosing.
* Female participants must not be breastfeeding.
* Men must agree to use a highly effective method of birth control with partners of childbearing potential during the study and for 1 month after completion of study dosing.
* Current or past smoking history >10 pack-years.
* Must be capable of performing reproducible spirometry maneuvers.

Exclusion Criteria:

* History of significant respiratory disease other than COPD, and/ or requires daily long-term oxygen therapy.
* Exacerbation of COPD, lung infection within 6 weeks prior to study.
* Start of or change in dose of COPD treatment 4 weeks before study.
* Daily using of maintenance systemic/inhaled corticosteroids (>1000 microgram of fluticasone propionate equivalent or >5 mg prednisone).
* Use of bronchodilators or medication for the treatment of COPD, aspirin, anti-inflammatories for a specific time, prior to the first dose or is not willing to abstain from their use for the specified time periods prior to study dose administration.
* Symptomatic prostrate hypertrophy, bladder neck obstruction, active cancer, narrow angle glaucoma.
* Clinical significant hypersensitivity to medications.
* Participants have an uncontrolled hematologic, immunologic, renal, neurologic, hepatic, endocrine or other disease that may place participant at risk.
* Cerebrovascular, cardiovascular disease or abnormal ECG.
* History of drug or alcohol abuse.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- P3 Research, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo A, Borin MT, Bourdet DL. Population Pharmacokinetics of Revefenacin in Patients with Chronic Obstructive Pulmonary Disease. Clin Pharmacokinet. 2021 Mar;60(3):391-401. doi: 10.1007/s40262-020-00938-3. PMID 33124005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21-May-2011 (FPFV) through 07-Oct-2011 (LPLV)
Pre-assignment Details: Male and female subjects between the ages of 40 and 75 years-old with a clinical diagnosis of COPD and responsiveness to ipratropium bromide.
Groups:
- Sequence 1: 1. Intervention 1 (Placebo) - [2 days], washout [7 days],
  2. Intervention 2 (TD4208 700 μg) - [2 days], washout [7 days],
  3. Intervention 3 (TD-4208 350 μg) - [2 days], washout [7 days],
  4. Intervention 4 (Ipratropium 500 μg) - [2 days], washout [7 days]
- Sequence 2: 1. Intervention 1 (TD-4208 700 μg) - [2 days], washout [7 days],
  2. Intervention 2 (Ipratropium 500 μg) - [2 days], washout [7 days],
  3. Intervention 3 (Placebo) - [2 days], washout [7 days],
  4. Intervention 4 (TD-4208 350 μg) - [2 days], washout [7 days]
- Sequence 3: 1. Intervention 1 (TD-4208 350 μg) - [2 days], washout [7 days],
  2. Intervention 2 (Placebo) - [2 days], washout [7 days],
  3. Intervention 3 (Ipratropium 500 μg) - [2 days], washout [7 days],
  4. Intervention 4 (TD-4208 700 μg) - [2 days], washout [7 days]
- Sequence 4: 1. Intervention 1(Ipratropium 500 μg) - [2 days], washout [7 days],
  2. Intervention 2 (TD-4208 350 μg) - [2 days], washout [7 days],
  3. Intervention 3 (TD-4208 700 μg) - [2 days], washout [7 days],
  4. Intervention 4 (Placebo) - [2 days], washout [7 days]
Period: Intervention 1 (2 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Intervention 2 (2 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Intervention 3 (2 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Intervention 4 (2 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: 1. Intervention 1 (Placebo) - [2 days], washout [7 days],
  2. Intervention 2 (TD-4208 700 μg) - [2 days], washout [7 days],
  3. Intervention 3 (TD-4208 350 μg) - [2 days], washout [7 days],
  4. Intervention 4 (Ipratropium 500 μg) - [2 days], washout [7 days]
- Sequence 4: 1. Intervention 1 (Ipratropium 500 μg) - [2 days], washout [7 days],
  2. Intervention 2 (TD-4208 350 μg) - [2 days], washout [7 days],
  3. Intervention 3 (TD-4208 700 μg) - [2 days], washout [7 days],
  4. Intervention 4 (Placebo) - [2 days], washout [7 days]
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 7 | 4 | 22
  >=65 years | 1 | 4 | 1 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.25 (7.48) | 63.25 (8.21) | 59.63 (3.67) | 64.88 (7.75) | 62.00 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 3 | 10
  Male | 5 | 6 | 6 | 5 | 22
Region of Enrollment [Number; unit: participants]
  New Zealand | 4 | 4 | 4 | 4 | 16
  South Africa | 4 | 4 | 4 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Peak Forced Expiratory Volume in One Second (FEV1) Relative to Baseline
Time Frame: From predose to 25 hours postdose
Measure: Least Squares Mean (Standard Error); unit: mL
Groups:
- Placebo: Single dose of placebo administered via nebulizer
- TD-4208 700 μg: Single dose of TD-4208 700 μg administered via nebulizer
- TD-4208 350 μg: Single dose of TD-4208 350 μg administered via nebulizer
- Ipratropium 500 μg: Single dose of Ipratropium 500 μg administered via nebulizer
Arm/Group | Placebo | TD-4208 700 μg | TD-4208 350 μg | Ipratropium 500 μg
Number analyzed (Participants) | 32 | 32 | 32 | 32
mL | 1708.0 (32.7) | 1877.3 (32.7) | 1881.8 (32.7) | 1883.6 (32.8)
Statistical Analysis 1: Comparison: Placebo vs TD-4208 350 μg; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 173.8, 95% CI 2-sided [112.4 to 235.3]
Statistical Analysis 2: Comparison: Placebo vs TD-4208 700 μg; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 169.3, 95% CI 2-sided [107.8 to 230.8]
Statistical Analysis 3: Comparison: Placebo vs Ipratropium 500 μg; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 175.6, 95% CI 2-sided [114.1 to 237.2]

2. Secondary Outcome: Area Under the FEV1 vs. Time Curve, Time-matched Difference From Placebo
Time Frame: 12 hr and 24 hr
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | TD-4208 700 μg | TD-4208 350 μg | Ipratropium 500 μg
Number analyzed (Participants) | 32 | 32 | 32 | 32
mL
  FEV1 at 12hr | 1519.2 (30.9) | 1642.6 (31.4) | 1631.7 (30.9) | 1534.5 (31.4)
  FEV1 at 24 hr | 1533.8 (22.4) | 1670.4 (22.4) | 1636.6 (22.4) | 1509.6 (22.4)
Statistical Analysis 1: Comparison: Placebo vs TD-4208 350 μg; Tx Difference of LS Mean FEV1 at 12 hr; Test type: Superiority; p = 0.001, t-test, 2 sided; Slope = 112.5, 95% CI 2-sided [44.5 to 180.5]
Statistical Analysis 2: Comparison: Placebo vs TD-4208 700 μg; Tx Difference of LS Mean FEV1 at 12 hr; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 123.4, 95% CI 2-sided [54.6 to 192.3]
Statistical Analysis 3: Comparison: Placebo vs Ipratropium 500 μg; Tx Difference of LS Mean FEV1 at 12 hr; Test type: Superiority; p = 0.659, t-test, 2 sided; Difference of LS Mean = 15.3, 95% CI 2-sided [-53.5 to 94.1]
Statistical Analysis 4: Comparison: Placebo vs TD-4208 350 μg; Tx Difference of LS Mean FEV1 at 24 hr; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 102.8, 95% CI 2-sided [54.1 to 151.5]
Statistical Analysis 5: Comparison: Placebo vs TD-4208 700 μg; Tx Difference of LS Mean FEV1 at 24 hr; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 136.6, 95% CI 2-sided [87.8 to 185.3]
Statistical Analysis 6: Comparison: Placebo vs Ipratropium 500 μg; Test type: Superiority — Tx Difference of LS Mean FEV1 at 24 hr; p = 0.327, t-test, 2 sided; Difference of LS Mean = -24.2, 95% CI 2-sided [-72.9 to 24.6]

3. Secondary Outcome: Area Under the FEV1 vs. Peak FEV1, Time-matched Difference From Placebo
Time Frame: 12 hr and 24 hr
Measure: Least Squares Mean (Standard Error); unit: hr*mL
Arm/Group | Placebo | TD-4208 700 μg | TD-4208 350 μg | Ipratropium 500 μg
Number analyzed (Participants) | 32 | 32 | 32 | 32
hr*mL
  AUC 0-12 hrs | 262.1 (4.2) | 291.2 (4.2) | 288.5 (4.2) | 287.7 (4.2)
  AUC 0-24 hrs | 261.2 (4.0) | 286.6 (4.0) | 281.3 (4.1) | 271.7 (4.0)
Statistical Analysis 1: Comparison: Placebo vs TD-4208 350 μg; Tx Difference of LS Mean AUC, 0-12 hrs; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 26.4, 95% CI 2-sided [18.0 to 34.8]
Statistical Analysis 2: Comparison: Placebo vs TD-4208 700 μg; Tx Difference of LS Mean AUC, 0-12 hrs; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 29.1, 95% CI 2-sided [20.8 to 37.4]
Statistical Analysis 3: Comparison: Placebo vs Ipratropium 500 μg; Tx Difference of LS Mean AUC, 0-12 hrs; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 25.6, 95% CI 2-sided [17.3 to 33.9]
Statistical Analysis 4: Comparison: Placebo vs TD-4208 350 μg; Tx Difference of LS Mean AUC, 0-24 hrs; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 20.1, 95% CI 2-sided [12.1 to 28.2]
Statistical Analysis 5: Comparison: Placebo vs TD-4208 700 μg; Tx Difference of LS Mean AUC, 0-24 hrs; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 25.4, 95% CI 2-sided [17.4 to 33.4]
Statistical Analysis 6: Comparison: Placebo vs Ipratropium 500 μg; Tx Difference of LS Mean AUC, 0-24 hr; Test type: Superiority; p = 0.010, t-test, 2 sided; Difference of LS Mean = 10.6, 95% CI 2-sided [2.5 to 18.6]

4. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) From 25% to 75% of Vital Capacity (FEF25-75), as Related to FEV1
Time Frame: 12hr and 24hr
Measure: Least Squares Mean (Standard Error); unit: L/sec
Arm/Group | Placebo | TD-4208 700 μg | TD-4208 350 μg | Ipratropium 500 μg
Number analyzed (Participants) | 32 | 32 | 32 | 32
L/sec
  Peak FEF 25-75% 24hr | 0.8 (0.0) | 0.9 (0.0) | 0.9 (0.0) | 0.9 (0.0)
  Peak FEF 25-75% 12hr | 0.8 (0.0) | 0.9 (0.0) | 0.9 (0.0) | 0.9 (0.0)
Statistical Analysis 1: Comparison: Placebo vs TD-4208 350 μg; Tx Difference of LS Mean 12 hr; Test type: Superiority; p = 0.003, t-test, 2 sided; Difference of LS Mean = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs TD-4208 700 μg; Tx Difference of LS Mean 12 hr; Test type: Superiority; p = 0.046, t-test, 2 sided; Difference of LS Mean = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs Ipratropium 500 μg; Tx Difference of LS Mean 12 hr; Test type: Superiority; p = 0.003, t-test, 2 sided; Difference of LS Mean = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 4: Comparison: Placebo vs TD-4208 350 μg; Tx Difference of LS Mean 24 hr; Test type: Superiority; p = 0.003, t-test, 2 sided; Difference of LS Mean = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 5: Comparison: Placebo vs TD-4208 700 μg; Tx Difference of LS Mean 24 hr; Test type: Superiority; p = 0.048, t-test, 2 sided; Difference of LS Mean = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 6: Comparison: Placebo vs Ipratropium 500 μg; Tx Difference of LS Mean 24 hr; Test type: Superiority; p = 0.007, t-test, 2 sided; Difference of LS Mean = 0.1, 95% CI 2-sided [0.0 to 0.2]

5. Secondary Outcome: Forced Expiratory Flow From 25% to 75% of Vital Capacity (FEF25-75), as Related to FEV1
Time Frame: 12hr and 24hr
Measure: Least Squares Mean (Standard Error); unit: L/sec
Arm/Group | Placebo | TD-4208 700 μg | TD-4208 350 μg | Ipratropium 500 μg
Number analyzed (Participants) | 32 | 31 | 32 | 31
L/sec
  FEF 25-75% at 12 hr | 0.6 (0.0) | 0.7 (0.0) | 0.7 (0.0) | 0.6 (0.0)
  FEF 25-75% at 24 hr | 0.6 (0.0) | 0.6 (0.0) | 0.6 (0.0) | 0.6 (0.0)
Statistical Analysis 1: Comparison: Placebo vs TD-4208 350 μg; Tx Difference of LS Mean 12 hr; Test type: Superiority; p = 0.054, t-test, 2 sided; Difference of LS Mean = 0.1, 95% CI 2-sided [-0.0 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs TD-4208 700 μg; Tx Difference of LS Mean 12 hr; Test type: Superiority; p = 0.045, t-test, 2 sided; Difference of LS Mean = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs Ipratropium 500 μg; Tx Difference of LS Mean 12 hr; Test type: Superiority; p = 0.503, t-test, 2 sided; Difference of LS Mean = 0.0, 95% CI 2-sided [-0.0 to 0.1]
Statistical Analysis 4: Comparison: Placebo vs TD-4208 350 μg; Tx Difference of LS Mean 24 hr; Test type: Superiority; p = 0.183, t-test, 2 sided; Difference of LS Mean = 0.0, 95% CI 2-sided [-0.0 to 0.1]
Statistical Analysis 5: Comparison: Placebo vs TD-4208 700 μg; Tx Difference of LS Mean 24 hr; Test type: Superiority; p = 0.422, t-test, 2 sided; Difference of LS Mean = 0.0, 95% CI 2-sided [-0.0 to 0.1]
Statistical Analysis 6: Comparison: Placebo vs Ipratropium 500 μg; Tx Difference of LS Mean 24 hr; Test type: Superiority; p = 0.287, t-test, 2 sided; Difference of LS Mean = 0.0, 95% CI 2-sided [-0.1 to 0.0]

6. Secondary Outcome: Forced Vital Capacity (FVC)
Time Frame: From predose to 25 hours postdose
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | TD-4208 700 μg | TD-4208 350 μg | Ipratropium 500 μg
Number analyzed (Participants) | 32 | 32 | 32 | 32
mL
  Predose | 2941.9 (771.4) | 2949.1 (623.5) | 2986.7 (800.8) | 2959.4 (696.7)
  15 min | 2873.4 (748.5) | 3166.9 (704.9) | 3119.3 (700.1) | 3339.7 (761.3)
  30 min | 2944.7 (718.8) | 3263.8 (676.2) | 3262.2 (810.1) | 3399.4 (789.5)
  45 min | 2927.2 (760.7) | 3324.7 (784.8) | 3328.8 (758.3) | 3394.1 (858.2)
  1 hour | 2968.1 (747.3) | 3269.4 (801.2) | 3361.9 (787.3) | 3379.4 (829.7)
  2 hours | 3062.5 (717.0) | 3363.1 (764.1) | 3408.8 (922.2) | 3441.6 (770.9)
  3 hours | 3122.2 (774.5) | 3430.4 (858.6) | 3420.3 (912.0) | 3474.1 (815.1)
  4 hours | 3177.8 (798.6) | 3386.3 (901.7) | 3340.9 (867.1) | 3368.8 (836.4)
  6 hours | 3192.6 (794.3) | 3442.8 (849.5) | 3220.6 (960.7) | 3295.3 (889.4)
  8 hours | 3197.2 (826.9) | 3259.4 (837.3) | 3301.6 (875.8) | 3305.2 (841.6)
  10 hours | 2958.7 (686.0) | 3335.3 (848.5) | 3339.4 (749.7) | 3180.3 (815.5)
  11 hours | 3156.2 (827.5) | 3296.2 (720.4) | 3295.5 (901.9) | 3162.3 (733.7)
  12 hours | 3092.8 (714.8) | 3229.4 (859.7) | 3265.1 (842.1) | 3131.3 (737.7)
  14 hours | 3114.4 (803.0) | 3333.1 (803.6) | 3319.1 (904.3) | 3123.8 (793.1)
  22 hours | 3033.8 (669.4) | 3314.5 (802.1) | 3147.2 (754.4) | 3010.0 (596.6)
  23 hours | 2999.7 (779.1) | 3349.4 (834.5) | 3232.2 (849.4) | 3006.3 (680.4)
  24 hours | 3018.1 (758.2) | 3345.6 (810.6) | 3243.1 (864.9) | 3031.6 (703.4)
  25 hours | 3172.8 (810.0) | 3392.5 (844.0) | 3295.2 (744.4) | 3219.4 (762.7)

7. Secondary Outcome: Area Under the Forced Vital Capacity (FVC) vs. Time Curve
Time Frame: 0-24 hours
Measure: Least Squares Mean (Standard Error); unit: hr*mL
Arm/Group | Placebo | TD-4208 700 μg | TD-4208 350 μg | Ipratropium 500 μg
Number analyzed (Participants) | 32 | 32 | 32 | 32
hr*mL | 74168.1 (1155.5) | 80057.0 (1155.3) | 78143.6 (1155.9) | 76822.7 (1155.2)
Statistical Analysis 1: Comparison: Placebo vs TD-4208 350 μg; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 3975.5, 95% CI 2-sided [2007.3 to 5943.7]
Statistical Analysis 2: Comparison: Placebo vs TD-4208 700 μg; Test type: Superiority; p < 0.001, t-test, 2 sided; Difference of LS Mean = 5888.9, 95% CI 2-sided [3924.4 to 7853.4]
Statistical Analysis 3: Comparison: Placebo vs Ipratropium 500 μg; Test type: Superiority; p = 0.009, t-test, 2 sided; Difference of LS Mean = 2654.7, 95% CI 2-sided [689.7 to 4619.6]

ADVERSE EVENTS:
Time Frame: 5 months (May-October 2011)
Arm/Group | Placebo | TD-4208 700 μg | TD-4208 350 μg | Ipratropium 500 μg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 10/32 | 6/32 | 4/32 | 7/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | TD-4208 700 μg (N=32) | TD-4208 350 μg (N=32) | Ipratropium 500 μg (N=32)
Headache (Nervous system disorders) | 6 (6) | 3 (3) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Electrocardiogram T Wave peaked (Investigations) | 1 (1) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may communicate the trial results generated by the PI, but only after the first publication or presentation of the combined study results generated by all participating sites. The Sponsor can then review trial results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.